CLINICAL TRIAL: NCT00029120
Title: MRI Contrast Imaging in the Evaluation and Follow-up of Patients With Memory Disorder and Healthy Controls
Brief Title: Evaluation of Age- and Alzheimer's Disease-Related Memory Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020095; 02-M-0095
Record Dates: First submitted 2002-01-05; First posted 2002-01-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-04-21

CONDITIONS: Alzheimer Disease; Dementia; Memory Disorder; Healthy
Keywords: Alzheimer's Disease; Spectroscopy; Longitudinal; Perfusion; Hippocampus; N-acetylaspartic Acid; Cerebral Blood Flow; Aging; Dementia; Alzheimer's; Memory Disorder; Memory; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders

SUMMARY:
The purpose of this study is to examine how a part of the brain called the hippocampus contributes to memory changes that occur with aging and Alzheimer's disease (AD).

Memory problems are the most important early symptoms of AD. The hippocampal region of the brain may be responsible for many age- and AD-related memory disorders. This study will use magnetic resonance imaging (MRI) scans to examine the structure, chemical composition, and function of the hippocampus in participants with AD, participants with mild memory problems, participants who are healthy but are at risk for AD, and healthy volunteers.

Participants in this study will undergo MRI scans of the brain. During the MRI, participants will perform memory tests to demonstrate hippocampal functioning.

DETAILED DESCRIPTION:
The major focus of the Geriatric Psychiatry Branch (GPB) is the study of individuals with memory disorders as a result of age or neurodegeneration. In particular, memory is the most important earliest clinical symptom of Alzheimer's disease (AD). Although the hippocampus may not be a biological determinant of all memories, there is a growing body of evidence suggesting that dysfunction of the hippocampus plays an important role in the most common forms of memory disorders. This proposal will allow for the application of an array of newly developed magnetic resonance imaging and spectroscopy methods to the study of hippocampal function in these patients. Most importantly, for the first time, structure, perfusion and neurochemical composition of the hippocampus in living individuals can be evaluated at high resolution without known risk. The study of longitudinal changes in hippocampal function should allow us to understand the contributions that various genotypes, e.g., ApoE4, and abnormalities in cerebrospinal fluid, e.g., A-beta42 and tau, play in the development of abnormal hippocampal structure and function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be referred through the GPB screening protocol 95-M-0096:

Subjects will include:

1. AD patients, diagnosis based on DSM-IV (APA Press, 1994) criteria,
2. Individuals over the age of 50 who are "at-risk" for AD on the basis of having first-degree relatives with AD and who tested within the normal range on a battery of cognitive tests at the time of initial inclusion,
3. Individuals with mild cognitive impairment (memory problems significant enough to concern the individual or members of the individual's family who do not meet the criteria for AD),
4. Control subjects, individuals without a positive family history of dementia in their first degree relatives and who test within the normal range on the battery of cognitive tests. As part of this screening process subjects who medical histories significant for any medical condition that would make it unsafe to perform MRI scans will be excluded.

EXLCUSION CRITERIA:

The same exclusion criteria used in those protocols for structural MRI and delineated under Hazards and Precautions would again be used.

All subjects participating in functional MRI scans will be required to be off prescription medications which could effect these scans, such as medications with anticholinergic effects, for two weeks-to one month prior to PET scan, and off psychotropic medication for one month. Withdrawal from psychotropic medications for purposes of participation in this protocol would only be considered for individuals already involved in the Longitudinal Study Protocol 95-M-0096.

Subjects will be cautioned not to consume alcohol, marijuana, or psychotropic drugs while on the study, nor to smoke, use caffeinated beverages, or take over-the counter medications such as cold medications (i.e.: benadryl, sudafed) for at least 12 hours prior to the functional MRI scans.

Pregnancy test will be conducted prior to MRI scans on women of childbearing age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2001-12-18; Study Completion 2008-04-21

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alvarez R, Alvarez V, Lahoz CH, Martinez C, Pena J, Sanchez JM, Guisasola LM, Salas-Puig J, Moris G, Vidal JA, Ribacoba R, Menes BB, Uria D, Coto E. Angiotensin converting enzyme and endothelial nitric oxide synthase DNA polymorphisms and late onset Alzheimer's disease. J Neurol Neurosurg Psychiatry. 1999 Dec;67(6):733-6. doi: 10.1136/jnnp.67.6.733. PMID 10567488